CLINICAL TRIAL: NCT01257269
Title: Thrombotic Thrombocytopenic Purpura Registry - A Prospective Observational Study for Patients Suffering From Hereditary Thrombotic Thrombocytopenic Purpura (Upshaw-Schulman Syndrome)
Brief Title: Genotype and Phenotype Correlation in Hereditary Thrombotic Thrombocytopenic Purpura (Upshaw-Schulman Syndrome)
Acronym: TTP registry
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Mach Gaensslen Foundation (Other); Baxalta Innovations GmbH, Wien, Austria (Unknown)
Responsible Party: Sponsor
Other Study IDs: 031/06
Record Dates: First submitted 2010-12-06; First posted 2010-12-09 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Thrombotic Thrombocytopenic Purpura; Congenital Thrombotic Thrombocytopenic Purpura; Familial Thrombotic Thrombocytopenic Purpura; Thrombotic Thrombocytopenic Purpura, Congenital; Upshaw-Schulman Syndrome
Keywords: Thrombotic thrombocytopenic purpura; ADAMTS13; Von Willebrand factor; Von Willebrand factor cleaving protease; Thrombocytopenia; Hemolytic anemia
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic; Thrombocytopenia; Anemia, Hemolytic | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with confirmed hereditary TTP due to congenital ADAMTS13 deficiency
  Interventions: Other: Observation
- 2: Family members of patients with confirmed hereditary TTP
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No interventions planned: treatment of patients at the discretion of the treating/responsible physician

SUMMARY:
Hereditary thrombotic thrombocytopenic purpura (Upshaw-Schulman syndrome) is a rare disorder characterized by thrombocytopenia as a result of platelet consumption, microangiopathic hemolytic anemia, occlusion of the microvasculature with von Willebrand factor-platelet-thrombic and ischemic end organ damage. The underlying patho-mechanism is a severe congenital ADAMTS13 (a disintegrin and metalloproteinase with thrombospondin type 1 motif, 13) deficiency which is the result of compound heterozygous or homozygous ADAMTS13 gene mutations.

Although considered a monogenic disorder the clinical presentation in Upshaw-Schulman syndrome patients varies considerably without an apparent genotype-phenotype correlation. In 2006 we have initiated a registry for patients with Upshaw-Schulman syndrome and their family members to identify possible triggers of acute bouts of TTP, to document individual clinical courses and treatment requirements as well as possible side effects of long standing plasma substitution, e.g. alloantibody formation or viral infections.

DETAILED DESCRIPTION:
Background

Thrombocytopenia and microangiopathic hemolytic anemia together with a severely deficient ADAMTS13 activity confirm the diagnosis of acute thrombotic thrombocytopenic purpura (TTP). Today two forms of classical TTP are distinguished. The acquired form is caused by circulating auto-antibodies, mainly Immunoglobulin G (IgG), inhibiting ADAMTS13 (a disintegrin and metalloproteinase with thrombospondin type 1 motif, 13) activity. In contrast, hereditary TTP, also known as Upshaw-Schulman syndrome (USS); #274150 Online Mendelian Inheritance in Man (OMIM), is the result of severe constitutional deficiency of ADAMTS13 due to compound heterozygous or homozygous mutations in the ADAMTS13 gene.

The clinical course of USS is variable with rather mild courses in some of the patients requiring plasma infusions only in special situations (i.e. pregnancy), while in others severe courses with important sequelae and even death in early childhood occur. The reasons for the variable clinical presentation and treatment requirements have not been elucidated. It seems likely, that additional, hitherto unidentified factors besides severe ADAMTS13 deficiency modify the clinical course.

At present, the clinical symptoms and laboratory values on which to base treatment regimens for hereditary TTP are poorly understood. Furthermore, increasing awareness of hereditary TTP results in rising numbers of patients in need of treatment and/or prophylaxis. However, currently very little is known on side effects of long standing plasma substitution. Alloimmunization with the formation of antibodies acting as inhibitors of treatment are well known in other congenital coagulation factor deficiencies (e.g. hemophilia A), but so far no case of treated hereditary TTP with subsequent antibody formation has been reported. It is the aim of the hereditary TTP Registry to provide information on the clinical course of the disease in as many patients as possible and therefore help to establish recommendations on the necessity, modalities, and risks of prophylactic plasma therapy in patients with hereditary TTP. Furthermore, it will help to gain detailed insight into triggers and risk factors of acute bouts of TTP.

Moreover, the hereditary TTP Registry will provide information for family members on their risk to develop TTP-like or TTP-related disorders.

Objective

Primary objective: Collection of as much information as possible on the clinical presentation, disease course, disease-modifying factors, and treatment modalities of patients suffering from hereditary thrombotic thrombocytopenic purpura (TTP).

Secondary objective: To document potential adversary effects of (long-term) plasma treatment in patients with hereditary thrombotic thrombocytopenic purpura (TTP).

Methods

The TTP Registry is designed to collect both retrospective and prospective clinical, molecular, and observational data on patients with confirmed or suspected hereditary TTP. Additionally, the Registry will collect data from family members of TTP patients enrolled in the Registry. The Registry will enroll as many confirmed or suspected hereditary TTP patients and their family members as possible; there is no cap on enrollment. The Registry enrollment and follow-up periods are open-ended. The endpoints for patients with confirmed or suspected hereditary TTP and family members are death or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Severe ADAMTS13 deficiency ( ≤ 10% activity) and no ADAMTS 13 inhibitor on two or more occasions at least one month apart
* Being a family member of a confirmed or suspected patient
* Molecular analysis of ADAMTS13 gene with one or more mutations and/or positive infusion trial (full recovered ADAMTS13 activity after infused fresh frozen plasma (FFP) with a plasma half-life of 2-4 days)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with either confirmed or with suspected hereditary TTP and their family members are eligible for enrollment
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2006-10; Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Clinical presentation and disease course in hereditary TTP | every year until death

SECONDARY OUTCOMES:
Identification of disease-modifying factors, including genotype-phenotype correlation | every year until death
Treatment requirements in hereditary TTP patients | every year until death
Documentation of potential adversary effects of (long-term) plasma treatment | every year until death
Mortality of hereditary TTP | every year until death
Clinical course in family members | every year until death

CONTACTS AND LOCATIONS:
Overall Officials: Johanna A Kremer Hovinga, MD, Study Chair — University Clinic of Hematology and Central Hematology Laboratory, Bern University Hospital and the University of Bern, Inselspital; Bernhard Lämmle, M.D., Study Chair — University Medical Center, Center for Thrombosis and Hemostasis, Mainz, Germany; Yoshihiro Fujimura, M.D., Study Chair — Department of Blood Transfusion Medicine, Nara Medical University, Kashihara, Japan; Ingrid Hrachovinova, Ph.D., Study Chair — Institute of Hematology and Blood Transfusion, Coagulation Laboratory, Prague, Czech Republic; Petter Quist-Paulsen, M.D., Ph.D., Study Chair — Department of Hematology, St Olavs Hospital, 7006 Trondheim, Norway; Reinhard Schneppenheim, M.D., Ph.D., Study Chair — Department of Pediatric Hematology and Oncology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany; James N. George, MD, Study Chair — University of Oklahoma Health Sciences Center, Department of Medicine, United States of America; Paul N Knoebl, MD, Study Chair — Medical University of Vienna, Div. Hematology and Hemostasis, Austria
Locations (7):
- University of Oklahoma Health Sciences Center, Department of Medicine, PO Box 26901, Oklahoma City, Oklahoma, United States
- Medical University of Vienna, Department of Medicine 1, Div. Hematology and Hemostasis Waehringer Guertel 18-20, Vienna, Austria
- Institute of Hematology and Blood Transfusion, Coagulation Laboratory, U nemocnice 1, Prague, Czechia
- University Medical Center Hamburg-Eppendorf, Department of Pediatric Hematology and Oncology, Martinistr 52, Hamburg, Germany
- Nara Medical University, Department of Blood Transfusion Medicine, Shijyo-cho 840, Kashihara, Nara, Japan
- Trondheim University St Olavs Hospital, Department of Hematology, PO Box 3250 Sluppen, Trondheim, Norway
- University Clinic of Hematology and Central Hematology Laboratory, Bern University Hospital and the University of Bern, Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Tarasco E, Butikofer L, Friedman KD, George JN, Hrachovinova I, Knobl PN, Matsumoto M, von Krogh AS, Aebi-Huber I, Cermakova Z, Gorska-Kosicka M, Jalowiec KA, Largiader CR, Prohaszka Z, Sinkovits G, Windyga J, Lammle B, Kremer Hovinga JA. Annual incidence and severity of acute episodes in hereditary thrombotic thrombocytopenic purpura. Blood. 2021 Jun 24;137(25):3563-3575. doi: 10.1182/blood.2020009801. PMID 33649760
- [Derived] van Dorland HA, Taleghani MM, Sakai K, Friedman KD, George JN, Hrachovinova I, Knobl PN, von Krogh AS, Schneppenheim R, Aebi-Huber I, Butikofer L, Largiader CR, Cermakova Z, Kokame K, Miyata T, Yagi H, Terrell DR, Vesely SK, Matsumoto M, Lammle B, Fujimura Y, Kremer Hovinga JA; Hereditary TTP Registry. The International Hereditary Thrombotic Thrombocytopenic Purpura Registry: key findings at enrollment until 2017. Haematologica. 2019 Oct;104(10):2107-2115. doi: 10.3324/haematol.2019.216796. Epub 2019 Feb 21. PMID 30792199
- [Derived] Fan X, Kremer Hovinga JA, Shirotani-Ikejima H, Eura Y, Hirai H, Honda S, Kokame K, Taleghani MM, von Krogh AS, Yoshida Y, Fujimura Y, Lammle B, Miyata T. Genetic variations in complement factors in patients with congenital thrombotic thrombocytopenic purpura with renal insufficiency. Int J Hematol. 2016 Mar;103(3):283-91. doi: 10.1007/s12185-015-1933-7. Epub 2016 Feb 1. PMID 26830967
- [Derived] Lammle B. VWF and complement. Blood. 2015 Feb 5;125(6):896-8. doi: 10.1182/blood-2014-12-612556. No abstract available. PMID 25655456
- [Derived] Mansouri Taleghani M, von Krogh AS, Fujimura Y, George JN, Hrachovinova I, Knobl PN, Quist-Paulsen P, Schneppenheim R, Lammle B, Kremer Hovinga JA. Hereditary thrombotic thrombocytopenic purpura and the hereditary TTP registry. Hamostaseologie. 2013 May 29;33(2):138-43. doi: 10.5482/HAMO-13-04-0026. PMID 23715103
- See also: Additional information — http://www.ttpregistry.net